CLINICAL TRIAL: NCT03223376
Title: A Phase III Study to Evaluate the Efficacy and Safety of Fruquintinib in Combination With Paclitaxel Versus Paclitaxel Alone in Second Line Gastric Cancer
Brief Title: A Phase III Study of Fruquintinib in Combination With Paclitaxel in Second Line Gastric Cancer(FRUTIGA)
Acronym: FRUTIGA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-013-00CH1
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fruquintinib+paclitaxel (Active Comparator): treatment arm (fruquintinib+paclitaxel) : Fruquintinib once daily, 3 weeks on/1week off combined with Paclitaxel 80mg/㎡ day1, 8, 15 of 4 weeks cycle.
  Interventions: Combination Product: fruquintinib +paclitaxel
- placebo+paclitaxel (Placebo Comparator): control arm (placebo+paclitaxel): Fruquintinib placebo once daily, 3 weeks on/1week off combined with Paclitaxel 80mg/㎡ day1, 8, 15 of 4 weeks cycle.
  Interventions: Combination Product: fruquintinib placebo + paclitaxel

INTERVENTIONS:
Combination Product: fruquintinib +paclitaxel — treatment arm(fruquintinib +paclitaxel)- subjects will receive Fruquintinib orally, once daily for 3 wks on/ 1 wk off combined with paclitaxel 80mg/㎡ at day 1,8,15 of 4-week cycle. Patients will receive a cycles of 4 weeks of study treatment or until the occurrence of progressive disease (PD), death, unacceptable toxicity, withdrawal of consent or other conditions that meet the end of treatment criteria.
  Other Names: HMPL-013+paclitaxel
  Arms: fruquintinib+paclitaxel
Combination Product: fruquintinib placebo + paclitaxel — control arm(fruquintinib placebo + paclitaxel)- subjects will receive Fruquintinib placebo orally, once daily for 3 wks on/ 1 wk off combined with paclitaxel 80mg/㎡ at day 1,8,15 of 4-week cycle. Patients will receive a cycles of 4 weeks of study treatment or until the occurrence of progressive disease (PD), death, unacceptable toxicity, withdrawal of consent or other conditions that meet the end of treatment criteria.
  Other Names: HMPL-013 placebo+paclitaxel
  Arms: placebo+paclitaxel

SUMMARY:
Fruquintinib once daily in 4 weeks treatment cycle (three weeks on and one week off) in combination with Paclitaxel 80mg/㎡（day1, 8, 15 of 4 weeks cycle) was well tolerated and demonstrated encouraging preliminary clinical antitumor activity in patients with advanced GC in ph1b/2 study. This study is aimed to evaluate the efficacy and safety of Fruquintinib in combination with Paclitaxel in the treatment of patients with aGC who have progressed after first line standard chemotherapy.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter Phase III clinical trial to compare the efficacy and safety of Fruquintinib combined with Paclitaxel versus Paclitaxel alone in patients with advanced gastric cancer who have progressed after first-line standard chemotherapy. After checking eligibility criteria, subjects will be randomized into Fruquintinib combined with Paclitaxel group (treatment group) or placebo combined with Paclitaxel group (control group) in a ratio of 1:1. Primary Efficacy Endpoint: Overall Survival (OS), Progression free survival (PFS) (According to RECIST Version 1.1). Secondary Efficacy Endpoints: Objective Response Rate (ORR), Disease Control Rate (DCR), Duration of Response (DOR), EORTC QLQ-C30 (V3) .Safety and tolerance will be evaluated by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 4.03.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Histologically or cytologically confirmed gastric or gastroesophageal junction adenocarcinoma
* Metastatic disease or locally advanced, unresectable disease
* Disease progression during or within 4 months after the last dose of the first-line therapy (with platinum/fluoropyrimidine )
* Adequate hepatic, renal, heart, and hematologic functions
* At least one measurable lesion (larger than 10 mm in diameter by spiral CT scan)
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure
* Good performance status Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 to 1

Exclusion Criteria:

* Pregnant or lactating women
* Any factors that influence the usage of oral administration
* Evidence of CNS metastasis
* Intercurrence with one of the following: non-controlled hypertension, coronary artery disease, arrhythmia and heart failure
* Abuse of alcohol or drugs
* Less than 4 weeks from the last clinical trial
* Previous treatment with VEGFR inhibition
* Disability of serious uncontrolled intercurrence infection
* Proteinuria ≥ 2+ (1.0g/24hr)
* Have evidence or a history of bleeding tendency within two months of the enrollment randomization, regardless of seriousness
* Within 12 months before the first treatment occurs artery/venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack) etc.
* Within 6 months before the first treatment occurs acute myocardial infarction, acute coronary syndrome or CABG
* Bone fracture or wounds that was not cured for a long time
* Coagulation dysfunction, hemorrhagic tendency or receiving anticoagulant Therapy
* The tumor invades a large vessel structure, such as the pulmonary artery, superior vena cava, or inferior vena cava

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 703 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | from randomization until death due to any cause, assessed up to 3 year
  every two months follow up after EOT observation period at 30 days after the last medication
Progression free survival (PFS) | from the date of randomization to the date of the first documented progressive disease or date of death due to any cause, assessed up to 1 year]
  PFS defined as the time from the date of randomization to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 1 year
  Tumor assessment will be performed using radiography method every 8 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Disease control rate (DCR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 1 year
  Tumor assessment will be performed using radiography method every 8 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Safety and tolerance evaluated by incidence, severity and outcomes of AEs | from first dose to 30 days post the last dose
  Safety and tolerance will be evaluated by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 4.03
Duration of response, DOR | : From the first documented PR or CR until the first documented PD or death，assessed up to 2 years
  DOR was the time from the date of first evidence of complete response or partial response to the date of objective progression or the date of death due to any cause, whichever is earlier. CR and PR were defined using the RECIST v1.1.
The European Organization for Reasearch and Treatment of Cancer（EORTC ） Quality of Life Questionnaire-Core 30 V3.0 (QLQ-C30 v3.0) | Evaluation before the beginning of each treatment cycle, at the end of treatment, and at the 30 days post the last dose，up to 2 years
  EORTC QLQ-C30 v3.0 was a self-administered questionnaire with multidimensional scales that measures global health status. There are 30 items in total, which can be divided into 15 fields. Five functional scales: physical function, role function, cognitive function, emotional function, social function; Three symptom scales: fatigue, pain, nausea and vomiting; Six individual measures: dyspnea, insomnia, loss of appetite, constipation, diarrhea, financial difficulties, and a global quality of life scale. The five functional scales and the global quality of life scale were scored independently. After linear transformation, the scores of all items ranged from 1 to 100, and the higher score, the higher functional level. The symptom scale was also scored independently and linearly transformed into a score from 1 to 100, with higher scores indicating more serious problems or symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, Principal Investigator — Sun Yat-sen University
Locations (7):
- China (7):
  - Hutchison Medi Pharma Invesigational sites, Hefei, Anhui
  - Hutchison Medi Pharma Investigational Site, Guangzhou, Guangdong
  - Hutchison Medi Pharma Investigational site, Harbin, Heilongjiang
  - Huchison Medi Pharma Investigational site, Nanjing, Jiangsu
  - Hutchison Medi Pharma Investigational sites, Hangzhou, Zhejiang
  - Hutchison Medi Pharma Investigational sites, Beijing
  - Hutchison Medi Pharma Investigational site, Shanghai

REFERENCES:
- [Derived] Wang F, Shen L, Guo W, Liu T, Li J, Qin S, Bai Y, Chen Z, Wang J, Pan Y, Shu Y, Zhao F, Cheng Y, Ye F, Gu K, Zhang T, Pan H, Zhong H, Zhou F, Qin Y, Yang L, Mao W, Li Q, Dai W, Li W, Wang S, Tang Y, Ma D, Yin X, Deng Y, Yuan Y, Li M, Hu W, Chen D, Li G, Liu Q, Tan P, Fan S, Shi M, Su W, Xu RH. Fruquintinib plus paclitaxel versus placebo plus paclitaxel for gastric or gastroesophageal junction adenocarcinoma: the randomized phase 3 FRUTIGA trial. Nat Med. 2024 Aug;30(8):2189-2198. doi: 10.1038/s41591-024-02989-6. Epub 2024 Jun 1. PMID 38824242